CLINICAL TRIAL: NCT00068731
Title: A Phase II Trial Of Lycopene For Patients With Asymptomatic Androgen-Independent Metastatic Prostate Cancer With PSA Elevation
Brief Title: Lycopene in Treating Patients With Metastatic Prostate Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCCTG-N0351; NCI-2012-02555 (Registry Identifier: CTRP (Clinical Trials Reporting System)); CDR0000327843 (Registry Identifier: PDQ (Physician Data Query))
Record Dates: First submitted 2003-09-10; First posted 2003-09-11 (Estimated); Last update posted 2016-07-13 (Estimated); Status verified 2016-07

CONDITIONS: Prostate Cancer
Keywords: stage IV prostate cancer; recurrent prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms | interventions — Lycopene

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- lycopene (Experimental): Patients receive oral lycopene twice daily on days 1-28. Courses repeat every 28 days for at least 4 months in the absence of disease progression or unacceptable toxicity.
  Patients are followed every 3 months until disease progression and then every 6 months for up to 5 years.
  Interventions: Dietary Supplement: lycopene

INTERVENTIONS:
Dietary Supplement: lycopene

SUMMARY:
RATIONALE: Lycopene, a substance found in tomatoes, may lower prostate-specific antigen (PSA) levels and slow or prevent the development of prostate cancer.

PURPOSE: Phase II trial to study the effectiveness of lycopene in treating patients who have asymptomatic metastatic prostate cancer and a rising PSA level.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine the percentage of patients with asymptomatic androgen-independent metastatic prostate cancer and an elevated prostate-specific antigen (PSA) level who sustain a decline in PSA after 4 months of treatment with lycopene.

Secondary

* Determine the response duration of PSA decline in patients treated with this therapy.
* Determine the time to the first consistent PSA increase in patients treated with this therapy.
* Determine whether a decline in PSA coincides with evidence of disease regression on physical examination or radiographic assessment in patients treated with this therapy.
* Determine the adverse event profile of this therapy in these patients.
* Determine the factors that motivate prostate cancer patients to enroll in a nutritional-based therapy study.

OUTLINE: This is a multicenter study.

Patients receive oral lycopene twice daily on days 1-28. Courses repeat every 28 days for at least 4 months in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 months until disease progression and then every 6 months for up to 5 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of androgen-independent prostate cancer
* Asymptomatic metastatic disease

  * Unlikely to become symptomatic within the next 4 months
  * No bone pain, shortness of breath, fatigue, or urinary symptoms directly attributable to prostate cancer
* Radiologic, physically palpable, and/or biochemical evidence of tumor progression after prior orchiectomy OR during treatment with a luteinizing hormone-releasing hormone (LHRH) agonist OR after initiation of another hormonal agent
* Sustained prostate-specific antigen (PSA) elevation, defined by the following:

  * PSA greater than 5 ng/mL
  * At least 2 consecutive increases in PSA at least 1 week apart
  * Sustained increase in PSA at least 4 weeks after discontinuation of prior flutamide (or other antiandrogen therapy) or megestrol AND at least 6 weeks after discontinuation of prior bicalutamide
* No known CNS metastases or carcinomatous meningitis

PATIENT CHARACTERISTICS:

Age

* 18 and over

Performance status

* ECOG 0-2

Life expectancy

* At least 12 weeks

Hematopoietic

* Not specified

Hepatic

* Bilirubin no greater than 1.5 mg/dL* NOTE: *Includes patients with liver involvement secondary to tumor

Renal

* See Disease Characteristics
* Creatinine no greater than 2 times upper limit of normal

Pulmonary

* See Disease Characteristics

Other

* No other malignancy within the past 5 years except basal cell skin cancer
* No medical or psychiatric condition that would preclude study participation

PRIOR CONCURRENT THERAPY:

Biologic therapy

* More than 4 weeks since prior immunotherapy

Chemotherapy

* More than 4 weeks since prior chemotherapy
* No concurrent chemotherapy

Endocrine therapy

* See Disease Characteristics
* More than 4 weeks since prior hormonal therapy (other than an LHRH agonist)
* No concurrent corticosteroids
* No concurrent progestational agents
* No concurrent new hormonal therapy

Radiotherapy

* No concurrent radiotherapy, including radiotherapy for new bone disease

Surgery

* See Disease Characteristics

Other

* More than 4 weeks since other prior anticancer therapy
* No other concurrent investigational anticancer agents
* No other concurrent alternative medicine therapies (e.g., saw palmetto or PC-SPES)

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2004-01; Primary Completion 2007-02 (Actual); Study Completion 2009-10 (Actual)

PRIMARY OUTCOMES:
percentage of patients with asymptomatic androgen-independent metastatic prostate cancer and an elevated prostate-specific antigen (PSA) level who sustain a decline in PSA after 4 months of treatment with lycopene | Up to 4 months

SECONDARY OUTCOMES:
response duration | Up to 5 years
time to the first consistent PSA increase | Up to 5 years
disease regression | Up to 5 years

CONTACTS AND LOCATIONS:
Overall Officials: Aminah Jatoi, MD, Study Chair — Mayo Clinic
Locations (18):
- United States (18):
  - CCOP - Mayo Clinic Scottsdale Oncology Program, Scottsdale, Arizona
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - CCOP - Atlanta Regional, Atlanta, Georgia
  - CCOP - Illinois Oncology Research Association, Peoria, Illinois
  - CCOP - Carle Cancer Center, Urbana, Illinois
  - CCOP - Cedar Rapids Oncology Project, Cedar Rapids, Iowa
  - CCOP - Iowa Oncology Research Association, Des Moines, Iowa
  - Siouxland Hematology-Oncology, Sioux City, Iowa
  - CCOP - Wichita, Wichita, Kansas
  - CCOP - Ochsner, New Orleans, Louisiana
  - CCOP - Duluth, Duluth, Minnesota
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - Coborn Cancer Center, Saint Cloud, Minnesota
  - CCOP - Metro-Minnesota, Saint Louis Park, Minnesota
  - Medcenter One Health System, Bismarck, North Dakota
  - CCOP - Dayton, Dayton, Ohio
  - CCOP - Upstate Carolina, Spartanburg, South Carolina
  - CCOP - Sioux Community Cancer Consortium, Sioux Falls, South Dakota

REFERENCES:
- [Result] Jatoi A, Burch P, Hillman D, Vanyo JM, Dakhil S, Nikcevich D, Rowland K, Morton R, Flynn PJ, Young C, Tan W; North Central Cancer Treatment Group. A tomato-based, lycopene-containing intervention for androgen-independent prostate cancer: results of a Phase II study from the North Central Cancer Treatment Group. Urology. 2007 Feb;69(2):289-94. doi: 10.1016/j.urology.2006.10.019. PMID 17320666